CLINICAL TRIAL: NCT00148421
Title: A Study of Darbepoetin Alfa Administered Once Every 2 Weeks (Q2W) Compared With Epoetin Alfa Administered Once Every Week (QW) for the Treatment of Anemia in Subjects With Non-myeloid Malignancies Receiving Multicycle Chemotherapy.
Brief Title: Study for the Treatment of Anemia in Patients With Non-myeloid Malignancies Receiving Multicycle Chemotherapy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20030125
Record Dates: First submitted 2005-06-30; First posted 2005-09-08 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Anemia
Keywords: Non-myeloid malignancy; Chemotherapy-induced anemia
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa; Epoetin Alfa

INTERVENTIONS:
Drug: Darbepoetin alfa and Epoetin alfa

SUMMARY:
Comparing two drugs to treat subjects with non-myeloid malignancies receiving multicycle chemotherapy.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effect of darbepoetin alfa and Epoetin alfa for the treatment of anemia in subjects with non-myeloid malignancies receiving multicycle chemotherapy.

ELIGIBILITY:
Inclusion Criteria: - Planned chemotherapy treatment - Anemia (hemoglobin concentration less than or equal to 11.0 g/dL) - Adequate renal and liver function - Subjects must provide written informed consent Exclusion Criteria: - Known history of seizure disorder - Known primary hematologic disorder causing anemia other than non-myeloid malignancies - Unstable / uncontrolled cardiac condition - Clinically significant inflammatory disease - Known positive test for HIV infection - Neutralizing antibodies to rHuEPO - Epoetin alfa or darbepoetin alfa therapy within 4 weeks before randomization - Received any investigational drug or device within 30 days before randomization - Pregnant or breast feeding - Not using adequate contraceptive precautions - Previously randomized into this study - Known hypersensitivity to recombinant mammalian-derived product - Concerns for subject's compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Reduced incidence of transfusions

SECONDARY OUTCOMES:
Change in hemoglobin concentration

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] 20030125 Study Group Trial; Glaspy J, Vadhan-Raj S, Patel R, Bosserman L, Hu E, Lloyd RE, Boccia RV, Tomita D, Rossi G. Randomized comparison of every-2-week darbepoetin alfa and weekly epoetin alfa for the treatment of chemotherapy-induced anemia: the 20030125 Study Group Trial. J Clin Oncol. 2006 May 20;24(15):2290-7. doi: 10.1200/JCO.2005.03.8570. PMID 16710026
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com